CLINICAL TRIAL: NCT00418795
Title: A Multi-centre, Double-blind, Randomized, Placebo-controlled, Parallel Group Trial, Investigating the Efficacy and Safety of Porphozym (Recombinant Human Porphobilinogen Deaminase) in the Treatment of Acute Attacks in AIP
Brief Title: Porphozym in the Treatment of Acute Attacks in AIP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zymenex A/S (Industry)
Organization: Chiesi Farmaceutici S.p.A. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: rhPBGD-02
Expanded Access: Available
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Acute Intermittent Porphyria
Keywords: Acute Intermittent Porphyria; treatment; Acute attack
MeSH Terms: conditions — Porphyria, Acute Intermittent

INTERVENTIONS:
Drug: recombinant human porphobilinogen deaminase (Porphozym)

SUMMARY:
A multi-centre, double-blind, randomized, placebo controlled, parallel group trial, investigating the efficacy and safety of Porphozym (recombinant human porphobilinogen deaminase)in the treatment of acute attacks in AIP.

DETAILED DESCRIPTION:
The primary objective is: To investigate the biochemical efficacy on plasma porphobilinogen (PBG) of Porphozy(recombinant human porphobilinogen deaminase) in subjects with Acute Intermittent Porphyria (AIP) during an attack and the clinical efficacy clinical efficacy of Porphozym™, being the change in pain from baseline to 24 hours after start of treatment. The correlation between the biochemical and clinical efficacy is investigated as well. Further the safety of Porphozym™ is evaluated.

After a screening period lasting as short as possible subjects enrolled in the trial will be randomized to treatment with either Porphozym™ or placebo. Treatment is given over 48 hours. After end of treatment, the subject enters the observation period, which lasts until the discharge from the hospital. Subjects are followed up with visits 14 and 28 days after end of treatment. Additional safety follow-up will be performed 2, 4 and 6 months after end of treatment. At least 36 Subjects will be enrolled in the trial.

The trial drug,is supplied by Zymenex A/S, Denmark in vials for reconstitution in water for injections (WFI).

At start of treatment a bolus injection iv is given to decrease PBG levels ot zero. This is followed by continuous iv infusion of the enzyme over the following 48 hours.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Confirmed diagnosis of AIP
* Previous attacks with PBG above the reference level of the laboratory AND exclusion of variegate porphyria (florescence emission of plasma samples is maximal at 626 nm in VP) AND exclusion of hereditary coproporphyria (HCP) (increased ratio of fecal coproporphyrin III to coproporphyrin I found in HCP)
* Acute attack of AIP verified by presence of abdominal and/or back and/or limb pain, diagnosed by the investigator as being caused by AIP
* Urine PBG above 6 mmol/mol creatinine (5 times upper reference level of the central laboratory)
* Male or female aged above 18 year

Exclusion criteria are:

* First acute attack in AIP
* Other reasons for abdominal and/or back and/or limb pain as judged by the investigator
* Therapy with human hemin within 7 days prior to administration of trial drug
* Treatment with any investigational drug within 4 weeks prior to this trial
* Known or suspected allergy to the trial product or related products
* Pregnant or breast-feeding women and women who intend to become pregnant prior to or during the trial
* Women of child-bearing potential who are not using acceptable methods of contraception (systemic contraception, IUD, barrier method or GnRH analogues)
* Previous documented renal impairment defined as above 150 mmol/L or 1.7 mg/dL serum creatinine, indicating a reduction in kidney function of 50% or more
* Any disease or condition that the investigator judges would interfere with the trial
* Previous randomization in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2003-06-11 (Actual); Primary Completion 2006-06-20 (Actual); Study Completion 2006-06-20 (Actual)

PRIMARY OUTCOMES:
Change in Plasma PBG

CONTACTS AND LOCATIONS:
Overall Officials: Christer Andersson, MD, Principal Investigator — Umeå University
Locations (1):
- Univercity Texas Medical Branch, Galveston, Texas, United States